CLINICAL TRIAL: NCT05448079
Title: The Effect of Sexual Counseling Given According to the PLISSIT Model on Sexual Functions, Marital Adjustment and Quality of Sexual Life of Postmenopausal Women
Brief Title: The Effect of Sexual Counseling Given According to the PLISSIT Model on FSFI, MAS and SQOL-F of Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Ayşe Sevim AKBAY KISA, Principal Investigator, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SuleymanDUAyşeAKBAYKISA-001
Record Dates: First submitted 2022-05-24; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Postmenopause; Sexual Function; Marital Relationship

STUDY DESIGN:
Intervention Model Description: The sample was divided into intervention and control groups sexual counseling based on the PLISSIT model
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sexual counseling intervention group according to the PLISSIT model (Experimental): Sexual counseling according to the PLISSIT model, randomized pretest-posttest
  Interventions: Other: Sexual counseling according to the PLISSIT model, randomized pretest-posttest
- control (Experimental): Non-counseling group
  Interventions: Other: Sexual counseling according to the PLISSIT model, randomized pretest-posttest

INTERVENTIONS:
Other: Sexual counseling according to the PLISSIT model, randomized pretest-posttest — experimental and control ,a randomized pretest-posttest study to examine

SUMMARY:
This study was conducted as a randomized pretest-posttest study to examine the effect of sexual counseling based on the PLISSIT model on post-menopausal women's sexual functions, marital adjustment and quality of sexual life. Sixty women (Experimental=30, Control=30) that applied to the menopause policlinic of a Women Diseases Training and Research Hospital were included in the study. Two women dropped out later, so the study was completed with 58 (Experimental=29, Control=29) women. Firstly, women were separated into two groups according to the cut-point of (26,55) in The Female Sexual Function Index (FSFI) (those who score 26,6 and above or 26,5 and below) and then these two groups were divided into intervention and control groups randomly. Data were collected with Descriptive Questions Form, Menopause Symptom Evaluation Scale (MRS), FSFI, Marital adjustment Scale (MAS) and Sexual Quality of Life Questionnaire Scale - Female Version (SQOL-F) between September 07, 2020 and March 26, 2021. The intervention group was given sexual counselling, prepared in line with the PLISSIT model, for three weeks, once a week and lasting approximately one hour. The effect of the counseling was tested twelve weeks after counseling was completed. Women in the control group were also interviewed twice concurrent with the intervention group; once when the counseling began and once during the last assessment. Women in the control group filled some data forms. After the study was completed, the counseling was also given to women who wanted it, in the control group. Frequency and percentage values, descriptive statistics, Fisher's Exact Test, Pearson Chi Square, t tests, for non-normally distributed data Mann Whitney U test and the Wilcoxon test were used for data analysis.

Keywords: Post-menopausal period, sexual counseling, PLISSIT model, nursing care

DETAILED DESCRIPTION:
Akbay-Kısa, A. S., The effect of sexual counseling given according to the PLISSIT model on sexual functions, marital adjustment and quality of sexual life of postmenopausal women. Hacettepe University Graduate School Health Sciences, Obstetrics and Gynecological Nursing Programme, Doctorate Thesis, Ankara, 2021. This study was conducted as a randomized pretest-posttest study to examine the effect of sexual counseling based on the PLISSIT model on post-menopausal women's sexual functions, marital adjustment and quality of sexual life. Sixty women (Experimental=30, Control=30) that applied to the menopause policlinic of a Women Diseases Training and Research Hospital were included in the study. Two women dropped out later, so the study was completed with 58 (Experimental=29, Control=29) women. Firstly, women were separated into two groups according to the cut-point of (26,55) in The Female Sexual Function Index (those who score 26,6 and above or 26,5 and below) and then these two groups were divided into intervention and control groups randomly. Data were collected with Descriptive Questions Form, The Female Sexual Function Index, Marital adjustment Scale and Sexual Quality of Life Questionnaire Scale - Female Version between September 07, 2020 and March 26, 2021. Women were asked to fill the demographic questions form and survey forms based on their own self-evaluations while they were accompanied by the researcher. The intervention group was given sexual counselling, prepared in line with the PLISSIT model, for three weeks, once a week and lasting approximately one hour. The effect of the counseling was tested twelve weeks after counseling was completed. Women in the control group were also interviewed twice concurrent with the intervention group; once when the counseling began and once during the last assessment. During those interviews, women in the control group filled some data forms. After the study was completed, the counseling was also given to women who wanted it, in the control group. Frequency and percentage values, descriptive statistics, Fisher's Exact Test, Pearson Chi Square, t tests, for non-normally distributed data Mann Whitney U test and the Wilcoxon test were used for data analysis.

Keywords: Post-menopausal period, sexual counseling, PLISSIT model, nursing care

ELIGIBILITY:
Inclusion Criteria:

1. Being in the first year of postmenopause,
2. Living with spouse/partner,
3. Having an active sex life,
4. Being able to speak, understand and read Turkish,
5. Entering menopause naturally,
6. Living within the borders of Ankara province,
7. Not having menopause at an early or late age (over 40 years and under 55 years old),
8. Not taking hormone replacement therapy,
9. Not using herbal treatment for menopause (containing estrogen),
10. Not having a type of cancer that may affect sexual function,
11. Not receiving chemotherapy / radiotherapy,
12. No health problems (Hypertension, Diabetes, Cardiovascular disease, Urinary incontinence),
13. Not having a mental illness and/or not using drugs (antipsychotic drugs, Spironolactone, etc.),
14. Not being diagnosed with COVID in the last month,
15. Not having a sexual dysfunction diagnosis / treatment history in himself or his partner,
16. Not getting sexual health counseling before.

Exclusion Criteria:

1. Receiving sexual health counseling from another consultant during the working period,
2. Desiring to leave the research at any stage of the research,
3. Failure to attend at least one of the sexual health counseling sessions,
4. Not participating in the post-test,
5. Getting a diagnosis of COVID.

Ages: 42 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Postmenopause, female
Enrollment: 58 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2020-12-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index | 28.09.2020- 02.04.2021. The research period for a participant takes approximately four months.
  Rosen et al [2000] developed this scale. It includes 19 items. Responses to some items range from 0 to 5 while others range from 1 to 5. The scores are summed up to create single Female Sexual Function Index score that ranges from 2 to 36. Higher scores mean better sexual functions.
Marital Adjustment Subscale | 28.09.2020- 02.04.2021. The research period for a participant takes approximately four months.
  It was developed by Locke and Wallace (1959) and consists of 15 items. The validity and reliability for Turkish translation was conducted by Kışlak-Tutarel (1999). The response range for the items are as the following: Item 1 = 0-6 points, Item 2 to 9 = 0-5 points, Items 10, 12, and 14 = 0-2 points, Items 11 and 13 = 0-3 points, and Item 15 = 0-2 points. The scale minimum value is 0 and maximum value is 58. Higher scores mean better marital adjustment.
The Sexual Quality Of Life-Female | 28.09.2020- 02.04.2021. The research period for a participant takes approximately four months.
  It was developed by Symonds et al (2005) and consists of 18 items. Items are scored from 0 to 5. The scale minimum value is 0 and maximum value is 90. Higher scores mean better sexual quality in a women's life.
Menopause Rating Scale | 28.09.2020- 02.04.2021. The research period for a participant takes approximately four months.
  It was developed by Schneider et al (1992) The Turkish validity and reliability study was carried by Gürkan (2005). The scale has a minimum value of 0 and a maximum value of 44. Higher scores mean more symptoms in menopause.

CONTACTS AND LOCATIONS:
Overall Officials: Gülten HÜ Koç, asst. prof., Study Director — Hacettepe University; Berna EH Dilbaz, professor, Study Chair — Etlik Hastanesi
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No